CLINICAL TRIAL: NCT06341673
Title: Impact of Transcutaneous Tibial Nerve Stimulation on Bladder Storage Symptoms and Quality of Life in People With Multiple Sclerosis- A Randomised Controlled Trial"
Brief Title: Impact of TTNS on Bladder Symptoms Among People With MS, A RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hawra Al-Dandan (Other)
Responsible Party: Sponsor-Investigator, Hawra Al-Dandan, Senior specialist, Imam Abdulrahman Bin Faisal University
Organization: Imam Abdulrahman Bin Faisal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2023-O3-442
Record Dates: First submitted 2024-03-06; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Overactive Bladder Syndrome
Keywords: Multiple Sclerosis; Overactive bladder; Bladder storage symptoms; Incontinence; Tibial nerve stimulation; Stimulation
MeSH Terms: conditions — Multiple Sclerosis; Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Randomized, sham-controlled, double blind study with 1:1 allocation ratio.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and those who undertake data input and data analysis will be blind to group allocation to reduce the risk of performance bias. A principal investigator and co-investigator will insert data into SPSS so that the researchers can analyse data without having access to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm: Transcutaneous Electrical Nerve Stimulation- Transcutaneous Tibial Nerve Stimulation (Active Comparator): Participants will useTENS to stimulate tibial nerve on the medial side of the foot for 6 weeks, a total of 18 sessions, three times weekly for 30 minutes per session. All TENS units will be programmed and locked by principal investigator to ensure fixed stimulation parameters are used among participants throughout the study intervention. The stimulation frequency will be set at 10 Hz with a pulse duration 200 μs. Participants will be advised to apply the stimulation in a supine position or supported sitting with extended legs to avoid compression of nerve roots at the knee joint. Participants will place the stimulation electrode, the negative electrode, between 5 and 10 cm above the medial malleolus and the positive electrode behind the left medial malleolus.
  Interventions: Device: Active Transcutaneous Electrical Nerve Stimulation (TENS)
- Sham arm: Transcutaneous Electrical Nerve Stimulation (Sham Comparator): Participants randomized to the sham group, will place the TENS on the lateral side of the foot, the negative electrode on the top of the foot just above the small toe for conduction and the positive electrode on the bottom of below the smallest toe to avoid the tibial nerve and relevant cutaneous nerves. The location of conduction electrode was chosen since this location is proved to be away from bladder, pelvic, or major organ nerve acupuncture pathway. Participants will be instructed to raise up the intensity until the first and slight tingling sensation on the sole of the foot or toe. The stimulation will be used for 6 weeks, a total of 18 sessions, three times weekly for 30 minutes per session.
  Interventions: Device: Sham Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Active Transcutaneous Electrical Nerve Stimulation (TENS) — For active group: TENS is to be used to stimulate tibial Nerve at medial aspect of the foot. The stimulation is proved by flexion of the big toe (motor response) and/or tingling sensation of ipsilateral sole of foot (sensory response) by raising the current amplitude, mA, intensity. Increasing the intensity above sensory threshold is recommended but should not be painful
  Arms: Active arm: Transcutaneous Electrical Nerve Stimulation- Transcutaneous Tibial Nerve Stimulation
Device: Sham Transcutaneous Electrical Nerve Stimulation (TENS) — TENS on the lateral side of the foot, the negative electrode on the top of the foot just above the small toe for conduction and the positive electrode on the bottom of below the smallest toe to avoid the tibial nerve and relevant cutaneous nerves. Participants will be instructed to raise up the intensity until the first and slight tingling sensation on the sole of the foot or toe
  Arms: Sham arm: Transcutaneous Electrical Nerve Stimulation

SUMMARY:
Background: Neurogenic lower urinary tract dysfunction is common among people with multiple sclerosis (MS). Recent studies showed that bladder storage symptoms are predominant among MS with a pooled prevalence of frequency at 73.45% followed by urgency at 63.87%. Transcutaneous tibial nerve stimulation (TTNS) is a non-invasive treatment to manage bladder storage symptoms; however, the effectiveness of TTNS is based on a small number of studies with the absence of high-quality evidence. This study aims to investigate the effectiveness of TTNS on bladder storage symptoms compared with sham TTNS among people with MS.Methods: The investigators will use a randomised sham controlled double blind study to explore the effectiveness of TTNS in the treatment of bladder storage symptoms in MS. the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) was followed to standardize the conduct and reporting of the current protocol. The recruitment plan is twofold: 1) Open recruitment for people with MS through King Fahd Hospital of the University communication channels; 2) people with any type of MS attending their routine appointments in MS clinic at King Fahd Hospital of the University, Al Khobar. The investigators will investigate the effectiveness of TTNS compared to sham TTNS on bladder storage symptoms and the effect on quality of life using ICIQ-OAB, ICIQ 3-day bladder diary, ICIQ-LUTS qol, and PSQI. Participant's perception of change post intervention will be evaluated using GPE. Outcomes will be measured at 0, 6 weeks and at 6 months post intervention. A sample size of 72 patients (36 in each group) is required to achieve 90% power with two-tailed tests at an alpha level of 0.05.

Conclusion: Multiple sclerosis is a long-term condition, and self-management is important. TTNS provide a safe, non-invasive intervention that can be administered at home. Should the trial determine that TTNS is effective compared to sham TTNS, the investigators will plan to integrate TTNS into standard clinical care pathways in MS.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic inflammatory disease of the central nervous system (CNS) mainly affects young individuals. The mechanism responsible for MS initiates with the formation of acute inflammatory lesions categorized by breakdown of the blood-brain barrier (BBB) that causes scattered lesions in the brain and spinal cord , and it is the leading cause of autonomic dysfunction MS is increasingly a universal disease reported by joint project of the Multiple Sclerosis International Federation and the World Health Organization report . MS is more common in females than males with gender distribution ratio of 2.7:1. Likewise, the female: male ratio appears to be 3:1 in most developed countries.

The International Continence Society defines neurogenic lower urinary tract dysfunction (NLUTD) as lower urinary tract symptoms following neurological disease. The range and severity of neurogenic bladder symptoms depend on the location of the neurologic lesions, with more definite symptoms in people with MS associated with lesions at the pontine micturition centre (PMC) causing bladder storage symptoms and/ or the supra sacral lesions resulting in both bladder storage and voiding symptoms accompanied with an increased post-void residual. According to ICS classification of lower urinary tract symptoms terminology, bladder storage symptoms are a combination of urinary frequency, urinary urgency, nocturia, with or without urge urinary incontinence. Recent publication showed that bladder storage symptoms are the predominant symptoms among people with MS with an estimated pooled prevalence of frequency at 73.45% followed by urgency at 63.87%.

Several studies have reported the negative impacts of NLUTD on quality of life (QoL) among MS population including psychological distress, sleep disturbances, barriers to engaging in physical and social activities and disturbances of daily living. Previous studies showed the relationship between sleep disturbances and urinary symptoms. Also, sleep disturbance is associated with more severe urinary incontinence and overactive bladder symptoms. However, to date no studies have investigated the association of bladder storage symptoms and sleep disturbances among PwMS and bladder storage system and the possible impact of TTNS on quality of sleep among PwMS and bladder storage symptoms. Early diagnosis and proper management are of utmost importance in preserving good QoL among people with MS and urinary symptoms.

Management of bladder storage symptoms for neurogenic bladder population comprise pharmacological and non-pharmacological interventions. According to European Association of Urology (EAU), pharmacologic interventions include antimuscarinic which is considered as a first line intervention and Intradetrusor onabotulinumtoxin A (BOTOX) injections as a second-line treatment intervention. Non-pharmacologic interventions include patient education, life style modifications, behavioural interventions, pelvic floor muscle training (PFMT), and/ or neuromodulations. Tibial nerve stimulation (TNS) is a form of neuromodulation used to inhibit overactivity of detrusor muscle by using either a needle electrode (percutaneous tibial nerve stimulation) (PTNS), or adhesive pads (transcutaneous tibial nerve stimulation) (TTNS).

A number of small-scale studies demonstrate that tibial nerve stimulation (TTNS) may be a promising management approach for bladder storage symptoms in non-neurogenic and neurogenic bladder populations with the need of high quality studies to assess the effectiveness of this intervention. The exact mechanism by which TNS potentially treats bladder control is not yet fully understood.

To date no randomized controlled trials (RCT's) have been identified that explore the impact of TTNS on bladder storage symptoms, activity limitations and participation restrictions in people with MS. RCT's are required to provide a strong evidence-base for using TTNS among neurogenic bladder storage symptoms in MS. Recent publication of single-arm feasibility study showed that TTNS is feasible, safe, and acceptable as a treatment of bladder storage symptoms among PwMS. Therefore, there is a need to conduct RCTs using standardized reporting of outcome measures administering, widely available and affordable device, the transcutaneous electrical nerve stimulation (TENS) unit. In the current study the investigators chose the sham comparator to assess the efficacy of TTNS on bladder storage symptoms in MS population. Sham intervention enable to reduce uncertainty regarding the causal relationship between an intervention and outcome, also it is suitable in the beginning phases of efficacy-exploratory research when it is still unknown whether the given treatment has any effect.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory (with or without assistive device)
* Aged ≥18 years old
* Able to understand spoken and written Arabic Language
* Self-reported with at least one bladder storage symptom such as urinary frequency urinary urgency, nocturia, with or without urge urinary incontinence
* Willing to give written informed consent
* Able to understand how to complete the study outcome measures

Exclusion Criteria:

People with MS will be excluded if they have one or more of the following criteria at randomization:

* Indwelling urethral catheter
* Indwelling suprapubic catheter
* Bladder malignancy
* Diabetic mellitus
* Pregnant women or plan to be pregnant during the study intervention
* Recent pelvic related surgery <1 year
* Pacemaker or other metallic internal devices
* Urinary tract infections (UTIs) during recruitment phase
* Unable to understand the instructions relating to operating the unit
* Having a bladder BOTOX-injection in the last 12-month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-04-28 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The International Consultation of Incontinence Questionnaire- Overactive Bladder (ICIQ- OAB) | 2 months
  Patient-completed questionnaire to measure urinary frequency, urgency, and nocturia. The total score ranges from 0 to 16 with higher values indicating increased symptom severity. Bother scales are not incorporated in the overall score.
3- day Bladder diary | 2 months
  Patient-completed diary for 72 hours. Number of episodes of urinary frequency, nocturia, and incontinence/ 72 hours will be calculated and compared from baseline with higher values indicating increased symptom severity.
Urinary sensation scale. | 2 months
  Number of urgency episodes and severity of urgency/72 hours will be calculated and compared from baseline. The total score ranges from 0 to 4 with higher values indicating increased symptom severity.

SECONDARY OUTCOMES:
The International Consultation of incontinence Questionnaire, Lower Urinary Tract Symptoms, Quality of life (ICIQ - LUTS,Qol) | 2 months
  Patient-completed questionnaire to measure the impact of urinary symptoms in quality of life. Overall scores ranges from19-76 with greater values indicating increased impact on quality of life. Bother scales are not incorporated in the overall score but indicate impact of individual symptoms for the patient
Pittsburgh Sleep Quality Index (PSQI)-item 6 | 2 months
  The item scored on a 0-3-point scale, where 0 = very good sleep quality and 3 = very bad sleep quality
Global Perceived Effect (GPE) Scale | 2 months
  Participant's perception of change post intervention will be assessed using a numeric scale from -5 to 5 with higher values indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Hawra AL Dandan, PhD, Principal Investigator — Imam Abdulrahman Bin Faisal University
Locations (1):
- King Fahd Hospital of the University, Khobar, Eastern Providence, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No